CLINICAL TRIAL: NCT01375946
Title: A Pharmacokinetic And Wearability Study of the Agile TCDS AG200-15 Following Weekly Application Under Various External Conditions in Healthy Female Volunteers
Brief Title: Pharmacokinetic Study Of AGILE AG200-15 After Weekly Application Under Various Conditions in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ATI-CL16
Record Dates: First submitted 2011-06-13; First posted 2011-06-20 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: Pharmacokinetic Profile (PK) and Safety; PK analysis of EE and LNG
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG200-15 location (Experimental): The subject will wear AG200-15 for 7 days and be exposed to one of 5 external conditions (normal, treadmill, cold water, whirlpool, dry sauna).
  Interventions: Drug: AG200-15

INTERVENTIONS:
Drug: AG200-15 — There will be three treatment periods. Subjects will be randomly assigned to one of the five conditions for the treatment period. The subject will be exposed daily to the condition assigned while wearing the patch. The study patch will be worn for a 7 day treatment period, followed by a 7 day washout period. The total duration of the study is 6 weeks.
  Other Names: transdermal contraceptive delivery system, patch

SUMMARY:
A study to evaluate pharmacokinetic profile, wearability and safety of AG200-15, transdermal delivery of levonorgestrel (LNG) and ethinyl estradiol (EE), under normal conditions and external conditions of heat, humidity, cold water and exercise.

DETAILED DESCRIPTION:
Normal conditions - average daily living activities, Dry Sauna - 10 minutes at 168.8 - 179.6 degrees Fahrenheit, Whirlpool - 10 minutes at 102.2 - 105.8 degrees Fahrenheit, Treadmill - 20 - 30 minutes at 60-80% max heart rate, Cold Water - 5 - 15 minutes at 71.6 degrees Fahrenheit.

There will be three treatment periods. Subjects will be randomly assigned to one of the five conditions for the treatment period. The subject will be exposed daily to the condition assigned while wearing the patch. The study patch will be worn for a 7 day treatment period, followed by a 7 day washout period. The total duration of the study is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, ages 18-45
* Body mass index (BMI)of ≥18 and less than or equal to 32, and weight ≥ 110 lbs.
* Willing to use a non-hormonal method of contraception if of childbearing potential, or have already undergone previous bilateral tubal ligation or hysterectomy
* Willing to refrain from use of alcohol and grapefruit juice from 48 hours prior to patch application until completion of each treatment period
* Willing to give informed consent to participate in study

Exclusion Criteria:

* Known or suspected pregnancy
* Breast-feeding or within 1 month after stopping breast-feeding
* Smokers
* Any disease that may worsen with hormonal treatment
* Hypersensitivity to transdermal preparations or sensitivity to surgical/medical tape

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, MPH, Study Director — Agile Therapeutics
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AG200-15 Condition (NDC): The subject will wear AG200-15 for 7 days and be exposed to normal (N), dry sauna (D) then cold water (C)conditions
- AG200-15 Condition (CNW): The subject will wear AG200-15 for 7 days and be exposed to cold water (C), normal (N) then whirlpool (W)conditions
- AG200-15 Condition (WTN): The subject will wear AG200-15 for 7 days and be exposed to whirlpool (W), treadmill (T) then normal (N)conditions
- AG200-15 Condition (NCD): The subject will wear AG200-15 for 7 days and be exposed to normal (N), cold water (C) then dry sauna (D)conditions
- AG200-15 Condition (DNT): The subject will wear AG200-15 for 7 days and be exposed to dry sauna (D), normal (N) then treadmill (T)conditions
- AG200-15 Condition (TWN): The subject will wear AG200-15 for 7 days and be exposed to treadmill (T), whirlpool (W) then normal (N) conditions
Period: Overall Study
Arm/Group | AG200-15 Condition (NDC) | AG200-15 Condition (CNW) | AG200-15 Condition (WTN) | AG200-15 Condition (NCD) | AG200-15 Condition (DNT) | AG200-15 Condition (TWN)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- AG200-15 Condition: The subject will wear AG200-15 for 7 days and be exposed to one of 5 external conditions (normal, treadmill, cold water, whirlpool, dry sauna).
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.13 (6.469)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) (0-168) Profile of Levonorgestrel (LNG)
Description: AUC(0-168) profile of LNG for each external condition including dry sauna, normal, whirlpool, cold water, and treadmill exercise. The blood sampling for the pharmacokinetic evaluations was performed at the following time points: 0 hour (immediately prior to dosing) and at 6 hours, 12 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days), 120 hours (5 days), 144 hours (6 days), and 168 hours (7 days) following application of the patch.
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
ng*hr/mL
  Normal | 157 (74)
  Dry Sauna: number analyzed (Participants) | 12
  Dry Sauna | 118 (51)
  Cold water: number analyzed (Participants) | 12
  Cold water | 153 (76)
  Whirlpool: number analyzed (Participants) | 12
  Whirlpool | 137 (81)
  Treadmill: number analyzed (Participants) | 12
  Treadmill | 119 (46)

2. Primary Outcome: AUC(0-168) Profile of Ethinyl Estradiol (EE)
Description: AUC(0-168) profile of EE for external condition including dry sauna, normal, whirlpool, cold water, and treadmill exercise. The blood sampling for the pharmacokinetic evaluations was performed at the following time points: 0 hour (immediately prior to dosing) and at 6 hours, 12 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days), 120 hours (5 days), 144 hours (6 days), and 168 hours (7 days) following application of the patch.
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
ng*hr/mL
  Normal | 4.7 (1.6)
  Dry sauna: number analyzed (Participants) | 12
  Dry sauna | 4.3 (2.0)
  Cold water: number analyzed (Participants) | 12
  Cold water | 4.9 (2.3)
  Whirlpool: number analyzed (Participants) | 12
  Whirlpool | 4.3 (1.4)
  Treadmill: number analyzed (Participants) | 12
  Treadmill | 3.9 (1.1)

3. Primary Outcome: Steady-state Concentration (Css) (48-168) Profile of LNG
Description: Css (48-168) profile of LNG for external condition including dry sauna, normal, whirlpool, cold water, and treadmill exercise. The blood sampling for the pharmacokinetic evaluations was performed at the following time points: 0 hour (immediately prior to dosing) and at 6 hours, 12 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days), 120 hours (5 days), 144 hours (6 days), and 168 hours (7 days) following application of the patch.
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
pg/mL
  Normal | 1068 (494)
  Dry Sauna: number analyzed (Participants) | 12
  Dry Sauna | 793 (317)
  Cold water: number analyzed (Participants) | 12
  Cold water | 1033 (518)
  Whirlpool: number analyzed (Participants) | 12
  Whirlpool | 918 (512)
  Treadmill: number analyzed (Participants) | 12
  Treadmill | 814 (333)

4. Primary Outcome: Css (48-168) Profile of EE
Description: Css (48-168) profile of EE for external condition including dry sauna, normal, whirlpool, cold water, and treadmill exercise. The blood sampling for the pharmacokinetic evaluations was performed at the following time points: 0 hour (immediately prior to dosing) and at 6 hours, 12 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days), 120 hours (5 days), 144 hours (6 days), and 168 hours (7 days) following application of the patch.
Time Frame: 6 weeks
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
pg/mL
  Normal | 30 (12)
  Dry Sauna: number analyzed (Participants) | 12
  Dry Sauna | 28 (13)
  Cold water: number analyzed (Participants) | 12
  Cold water | 29 (14)
  Whirlpool: number analyzed (Participants) | 12
  Whirlpool | 27 (9)
  Treadmill: number analyzed (Participants) | 12
  Treadmill | 24 (8)

5. Secondary Outcome: Patch Adhesion
Description: Patch adhesion scores by investigator evaluation by external condition; including dry sauna, whirlpool, treadmill exercise, normal, and cold water conditions; using the following scale:
  0: >90% adhered (essentially no lift off of the skin)
  1. >75% adhered but <90% (some edges showing lift)
  2. >50% adhered but <75% (half of system lifts off)
  3. <50% (> half of system lifts off, but undetached)
  4. patch completely detached
  Patches were assessed prior to patch removal.
Time Frame: 6 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15 Condition
Number analyzed (Participants) | 24
Score
  Normal | 0.08 (0.282)
  Dry Sauna: number analyzed (Participants) | 12
  Dry Sauna | 0.08 (0.289)
  Cold water: number analyzed (Participants) | 12
  Cold water | 0 (0)
  Whirlpool: number analyzed (Participants) | 12
  Whirlpool | 0 (0)
  Treadmill: number analyzed (Participants) | 12
  Treadmill | 0.17 (0.577)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | AG200-15 Condition
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 23/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 Condition (N=24)
Gastrointestinal disorders (Gastrointestinal disorders) | 12 (12)
General disorders and administration site conditions (General disorders) | 13 (13)
Infections and infestations (Infections and infestations) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (4)
Nervous system disorders (Nervous system disorders) | 14 (14)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 16 (16)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL16 study is required prior to publication submission.